CLINICAL TRIAL: NCT03025282
Title: Exploratory Study to Evaluate the Safety and Efficacy of CD10367 in Subjects With Psoriasis
Brief Title: Safety and Efficacy of CD10367 in Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.112075; 2016-002774-12 (EudraCT Number)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Betamethasone Valerate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- CD10367 3% Solution - Non-desquamated zone (Experimental)
  Interventions: Drug: CD10367 3% Solution - Non-desquamated zone
- CD10367 1% Solution - Non-desquamated zone (Experimental)
  Interventions: Drug: CD10367 1% Solution - Non-desquamated zone
- CD10367 solution placebo - Non-desquamated zone (Placebo Comparator): CD10367 solution placebo serves as negative control.
  Interventions: Drug: CD10367 solution placebo - Non-desquamated zone
- Betneval ointment - Non-desquamated zone (Active Comparator): This comparator containing Betamethasone valerate 0.1% serves as positive control.
  Interventions: Drug: Betneval ointment - Non-desquamated zone
- CD10367 3% Solution - Desquamated zone (Experimental)
  Interventions: Drug: CD10367 3% Solution - Desquamated zone
- CD10367 solution placebo - Desquamated zone (Placebo Comparator)
  Interventions: Drug: CD10367 solution placebo - Desquamated zone

INTERVENTIONS:
Drug: CD10367 3% Solution - Non-desquamated zone — Once daily application for 3 weeks
  Arms: CD10367 3% Solution - Non-desquamated zone
Drug: CD10367 1% Solution - Non-desquamated zone — Once daily application for 3 weeks
  Arms: CD10367 1% Solution - Non-desquamated zone
Drug: CD10367 solution placebo - Non-desquamated zone — Once daily application for 3 weeks
  Arms: CD10367 solution placebo - Non-desquamated zone
Drug: Betneval ointment - Non-desquamated zone — Once daily application for 3 weeks
  Other Names: Betamethasone Valerate
  Arms: Betneval ointment - Non-desquamated zone
Drug: CD10367 3% Solution - Desquamated zone — Once daily application for 3 weeks
  Arms: CD10367 3% Solution - Desquamated zone
Drug: CD10367 solution placebo - Desquamated zone — Once daily application for 3 weeks
  Arms: CD10367 solution placebo - Desquamated zone

SUMMARY:
This was an exploratory, single-center, investigator blinded, randomized, controlled, intra-individual study, involving participants with psoriasis vulgaris.

The objective was to evaluate, in a modified Dumas-Scholtz psoriasis mini-zone test, the safety and efficacy of CD10367 solution at 1% and 3% after a 3-week treatment period of once daily application.

DETAILED DESCRIPTION:
Study drugs would be applied in each participant once daily, 5 days a week during the first 2 weeks and for 4 days the third week on 6 mini-zones located on at least 2 psoriatic plaques as described below:

* on 2 mini-zones pretreated by a keratolytic product, would be tested:

  * CD10367 3% solution
  * CD10367 solution placebo
* on 4 mini-zones non-pretreated, would be tested:

  * CD10367 3% solution
  * CD10367 1% solution
  * CD10367 solution placebo
  * Betneval 0.1% ointment

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female aged at least 18 and up to 70 years old inclusive at screening visit.
2. Female of non childbearing potential (postmenopausal [absence of menstrual bleeding for 1 year prior to screening, without any other medical reason], hysterectomy or bilateral oophorectomy).
3. Participant had a skin phototype I to IV on Fitzpatrick's scale. (Screening visit).
4. The participant had a clinical diagnosis of stable plaque psoriasis, defined as no flare during the month before Screening visit and no change between Screening visit and Baseline visit, of mild to moderate severity. (Screening visit and Baseline Visit).
5. The participant presented with at least six eligible mini-zones, on at least two psoriasis plaques (Screening visit and verified also at Baseline Visit) with specific severity grades,
6. Participant agreed not to wear his/her contact lenses from the Baseline visit till the D19 visit (Screening visit).

Exclusion Criteria:

1. The participant presented guttate, erythrodermic, exfoliative, inverse, pustular, palmo plantar, infected or ulcerated psoriasis (Screening visit).
2. The participant had any uncontrolled or serious disease, or any medical or surgical condition, that might either interfere with the interpretation of the clinical trial results, and/or put the participant at significant risk (according to Investigator's judgment) if he/she participated in the clinical trial (e.g. history of on-going gastric or duodenal ulcer, clinically significant lung disease, etc.) (Screening visit).
3. The participant had known or suspected allergies or sensitivities to any components of the study drugs or of the keratolytic product (see Investigator's Brochure/Product label). (Screening visit).
4. The participant had known history of adverse drug reaction or hypersensitivity to a product with the same mode of action.
5. The participant had any abnormal clinically significant findings according to the ophthalmologist, at the ophthalmological exam at Screening visit,
6. The participant presented any abnormal laboratory tests judged clinically significant by the investigator (blood samplings and urinalysis done at Screening visit),
7. The participant had QTc interval >450 millisecond (msec) or any abnormal electrocardiogram (ECG) value considered as clinically significant by the cardiologist (Screening visit).
8. The participant had received, applied or taken some specified treatments within the specified time frame prior to the Baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Galderma Investigational Site, Nice, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in France from 03-November-2016 to 24-March-2017.
Pre-assignment Details: A total of 29 participants were screened, of which 24 participants were enrolled and randomized to receive the study treatments on 6 target mini-zones (on upper and/or the lower extremities [elbows, knees and tibiae shin area excluded] and/or on the trunk).
Units Other Than Participants: mini-zones
Groups:
- All Participants: Participants received 50 microliter (mcL) of 3 percent (3%) CD10367 solution and their matched placebo topically, on one or two desquamated psoriatic plaque (pre-treated) and 50 mcL of 3%, 1% CD10367 solution, their matched placebo and Betneval® 0.1% (positive control) topically, on one or two non-desquamated psoriatic plaque once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
Period: Overall Study
Arm/Group | All Participants
Started | 24; 144 mini-zones
Completed | 24; 144 mini-zones
Not Completed | 0; 0 mini-zones

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat (ITT) population that included all randomized participants.
Groups:
- All Participants: Participants received 50 mcL of 3% CD10367 solution or their matched placebo topically, on one or two desquamated psoriatic plaque (pre-treated) and 50 mcL of 3% and 1% CD10367 solution or their matched placebo and Betneval® 0.1% (positive control) topically, on one or two non-desquamated psoriatic plaque (pre-treated) once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Total Sum Score (Sum of Erythema, Scaling and Induration Scores)
Description: The TSS is the sum of the individual clinical scores of erythema, scaling and induration determined on a mini-zone. Each score was evaluated by the Investigator on all mini-zones using a 5-point scale (0: none; 1: mild; 2: moderate; 3: severe; 4: very severe) and were summed to obtain the Total Sum Score (TSS). Maximum total score was 12 (very severe); minimum total score was 0 (None). The mean AUC of TSSs were calculated for each intervention for all participants.
Time Frame: Day 1 to Day 19
Population: Analysis was performed on ITT population, which comprised of all participants who were randomized
Measure: Mean (Standard Deviation); unit: score on a scale*days
Units Other Than Participants: mini-zones
Groups:
- CD10367 Placebo Pretreated: Participants received 50 mcL of matched placebo solution topically, on one or two desquamated psoriatic plaque (pre-treated), once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 3% Pretreated: Participants received 50 mcL of 3% CD10367 solution topically, on one or two desquamated psoriatic plaque (pre-treated), once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 Placebo: Participants received 50 mcL of matched placebo solution topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 1%: Participants received 50 mcL of 1% CD10367 solution topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 3%: Participants received 50 mcL of 3% CD10367 solution topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- Betneval 0.1%: Participants received 50 mcL of 0.1% Betneval ointment topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale*days | 103.4 (24.5) | 101.7 (22.5) | 118.0 (23.2) | 118.6 (24.0) | 116.6 (26.3) | 75.3 (16.3)

2. Secondary Outcome: Area Under the Curve (AUC) of Individual Clinical Scores
Description: Each mini zone was evaluated by recording individual clinical scores (items: erythema, scaling, induration) for each participant using 5-point scale for each item and score ranged from 0(none), 1(mild), 2(moderate), 3(severe) and 4(very severe). Erythema: 0=No detectable erythema,1=Slight pinkness present, 2=Definite redness, easily recognized, 3=Intense redness, 4=Very intense redness; Scaling: 0=No shedding, 1=Barely perceptible shedding, noticeable only on light scratching or rubbing, 2=Obvious but not profuse shedding, 3=Heavy scale production, 4=Very thick scales; Induration: 0=Normal skin thickness/No elevation of skin, 1=Barely perceptible elevation (by touching) of the psoriasis plaques, 2=Obvious elevation above normal skin level/moderate thickening, 3=Definite thick elevation above normal skin level, 4=Very thick elevation. Higher score indicated worst conditions. The mean AUC for each intervention was calculated for each participant.
Time Frame: Day 1 to Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized
Measure: Mean (Standard Deviation); unit: score on a scale*days
Units Other Than Participants: mini-zones
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale*days
  Erythema | 37.1 (7.7) | 37.7 (7.6) | 42.7 (7.5) | 41.3 (7.7) | 41.7 (8.6) | 27.2 (7.4)
  Scaling | 32.3 (12.8) | 31.1 (11.3) | 38.4 (11.0) | 40.2 (11.8) | 39.6 (12.6) | 20.5 (4.9)
  Induration | 34.0 (5.6) | 32.9 (6.2) | 36.9 (7.2) | 37.1 (7.0) | 35.3 (7.8) | 27.5 (5.8)

3. Secondary Outcome: Total Sum Score (TSS) of Individual Clinical Scores
Description: The TSS was the sum of the individual clinical scores of erythema, scaling and induration determined on a mini-zone. Each score was evaluated by the Investigator on all mini-zones using a 5-point scale (0: none; 1: mild; 2: moderate; 3: severe; 4: very severe) and were summed to obtain the Total Sum Score (TSS). where maximum total score was 12 (worst condition) and minimum total score was 0 (no symptoms).
Time Frame: Day 1, Day 4, Day 8, Day 11, Day 15 and Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: mini-zones
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
score on a scale
  Day 1 | 5.0 (0.3) | 5.0 (0.3) | 7.3 (1.0) | 7.3 (1.0) | 7.3 (1.0) | 7.2 (1.0)
  Day 4 | 5.5 (1.1) | 5.6 (1.3) | 6.8 (1.3) | 6.7 (1.4) | 6.8 (1.3) | 4.5 (1.2)
  Day 8 | 6.4 (1.4) | 6.2 (1.4) | 7.1 (1.3) | 6.8 (1.8) | 6.8 (1.9) | 4.5 (1.1)
  Day 11 | 5.8 (1.6) | 5.8 (1.8) | 6.0 (1.7) | 6.4 (1.8) | 6.1 (2.1) | 3.5 (1.1)
  Day 15 | 5.9 (2.1) | 5.8 (1.8) | 6.5 (1.9) | 6.7 (1.6) | 6.5 (1.6) | 3.7 (1.2)
  Day 19 | 5.2 (2.3) | 4.8 (1.5) | 5.7 (1.5) | 5.7 (1.7) | 5.5 (1.9) | 3.0 (1.3)

4. Secondary Outcome: Percent Change in Total Sum Score (TSS)
Description: The TSS was the sum of the individual clinical scores of erythema, scaling and induration determined on a mini-zone. Each score was evaluated by the Investigator on all mini-zones using a 5-point scale (0: none; 1: mild; 2: moderate; 3: severe; 4: very severe) and were summed to obtain the Total Sum Score (TSS). where maximum score was 12 (worst condition) and minimum score was 0 (no symptoms). The TSS percentage change from Day 1 at each visit and erythema, scaling and induration scores and their changes from Day 1 at each visit were evaluated by visit and by treatment received.
Time Frame: Day 1, Day 4, Day 8, Day 11, Day 15 and Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized.
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: mini-zones
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
percent change
  Day 4 | 9.7 (20.0) | 11.6 (24.1) | -7.3 (11.4) | -7.4 (14.7) | -7.8 (13.0) | -36.6 (13.3)
  Day 8 | 28.3 (26.8) | 24.1 (25.5) | -2.9 (11.0) | -6.1 (17.7) | -8.5 (20.6) | -36.9 (14.1)
  Day 11 | 15.0 (30.6) | 16.1 (32.2) | -17.4 (20.3) | -12.2 (21.2) | -17.0 (22.7) | -51.9 (13.2)
  Day 15 | 17.6 (38.5) | 14.4 (31.4) | -11.7 (21.9) | -7.4 (21.4) | -11.7 (17.2) | -48.1 (14.9)
  Day 19 | 3.4 (43.3) | -5.8 (25.5) | -22.3 (18.0) | -22.0 (19.4) | -26.6 (19.1) | -58.4 (16.6)

5. Secondary Outcome: Erythema, Scaling and Induration Scores at Each Visit
Description: Status of psoriasis for each mini zone was evaluated by recording individual clinical scores (items: erythema, scaling, induration) using 5-point scale for each item and score ranged from 0(none), 1(mild), 2(moderate), 3(severe) and 4(very severe). Erythema: 0=No detectable erythema,1=Slight pinkness present, 2=Definite redness, easily recognized, 3=Intense redness, 4=Very intense redness; Scaling: 0=No shedding, 1=Barely perceptible shedding, noticeable only on light scratching or rubbing, 2=Obvious but not profuse shedding, 3=Heavy scale production, 4=Very thick scales; Induration: 0=Normal skin thickness/No elevation of skin, 1=Barely perceptible elevation (by touching) of the psoriasis plaques, 2=Obvious elevation above normal skin level/moderate thickening, 3=Definite thick elevation above normal skin level, 4=Very thick elevation. Higher score indicated worst conditions.
Time Frame: Day 1, Day 4, Day 8, Day 11, Day 15 and Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized
Measure: Mean (Standard Deviation); unit: score on scale
Units Other Than Participants: mini-zones
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
score on scale
  Erythema: Day 1 | 2.0 (0.2) | 2.0 (0.2) | 2.6 (0.5) | 2.5 (0.5) | 2.6 (0.5) | 2.5 (0.5)
  Erythema: Day 4 | 2.0 (0.4) | 2.1 (0.5) | 2.5 (0.6) | 2.4 (0.7) | 2.3 (0.6) | 1.5 (0.6)
  Erythema: Day 8 | 2.3 (0.6) | 2.3 (0.5) | 2.5 (0.6) | 2.3 (0.6) | 2.4 (0.7) | 1.5 (0.5)
  Erythema: Day 11 | 2.0 (0.5) | 2.1 (0.6) | 2.3 (0.5) | 2.2 (0.7) | 2.2 (0.7) | 1.3 (0.5)
  Erythema: Day 15 | 2.0 (0.7) | 2.1 (0.6) | 2.3 (0.6) | 2.3 (0.5) | 2.4 (0.6) | 1.4 (0.6)
  Erythema: Day 19 | 1.9 (0.7) | 1.8 (0.5) | 2.0 (0.6) | 2.1 (0.4) | 2.0 (0.6) | 1.1 (0.5)
  Scaling: Day 1 | 1.0 (0.2) | 1.0 (0.2) | 2.5 (0.5) | 2.5 (0.5) | 2.6 (0.5) | 2.5 (0.5)
  Scaling: Day 4 | 1.5 (0.7) | 1.5 (0.8) | 2.2 (0.6) | 2.3 (0.7) | 2.4 (0.6) | 1.2 (0.5)
  Scaling: Day 8 | 2.1 (0.8) | 2.0 (0.8) | 2.4 (0.7) | 2.3 (0.9) | 2.3 (1.0) | 1.3 (0.4)
  Scaling: Day 11 | 1.9 (0.9) | 2.0 (0.9) | 2.0 (0.8) | 2.2 (0.9) | 2.1 (1.1) | 0.8 (0.5)
  Scaling: Day 15 | 2.0 (1.0) | 1.8 (0.9) | 2.0 (0.9) | 2.3 (0.9) | 2.1 (0.9) | 1.0 (0.4)
  Scaling: Day 19 | 1.7 (1.0) | 1.4 (0.6) | 1.7 (0.8) | 1.7 (1.0) | 1.7 (0.8) | 0.7 (0.5)
  Induration: Day 1 | 2.0 (0.0) | 2.0 (0.0) | 2.2 (0.4) | 2.2 (0.4) | 2.1 (0.3) | 2.1 (0.3)
  Induration: Day 4 | 2.0 (0.2) | 1.9 (0.3) | 2.1 (0.3) | 2.0 (0.4) | 2.1 (0.4) | 1.8 (0.4)
  Induration: Day 8 | 2.0 (0.3) | 1.9 (0.4) | 2.2 (0.4) | 2.2 (0.5) | 2.0 (0.6) | 1.7 (0.5)
  Induration: Day 11 | 1.8 (0.5) | 1.7 (0.6) | 1.8 (0.6) | 2.0 (0.6) | 1.8 (0.7) | 1.3 (0.5)
  Induration: Day 15 | 1.9 (0.6) | 1.8 (0.6) | 2.1 (0.6) | 2.1 (0.5) | 2.0 (0.6) | 1.3 (0.5)
  Induration: Day 19 | 1.6 (0.8) | 1.6 (0.6) | 1.9 (0.5) | 1.9 (0.5) | 1.8 (0.7) | 1.1 (0.5)

6. Secondary Outcome: Percent Changes of Erythema, Scaling and Induration From Day 1 to Day 19
Description: as for outcome 5
Time Frame: Day 1, Day 4, Day 8, Day 11, Day 15, Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: mini-zones
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
percent change
  Erythema: Day 4 | -0.0 (0.4) | 0.1 (0.5) | -0.1 (0.4) | -0.1 (0.4) | -3.0 (0.5) | -1.0 (0.6)
  Erythema: Day 8 | 0.3 (0.5) | 0.2 (0.5) | -0.1 (0.4) | -0.2 (0.5) | -0.2 (0.6) | -1.0 (0.4)
  Erythema: Day 11 | 0.0 (0.4) | 0.1 (0.6) | -0.4 (0.7) | -0.3 (0.8) | -0.4 (0.8) | -1.2 (0.6)
  Erythema: Day 15 | -0.0 (0.6) | -0.0 (0.6) | -0.3 (0.7) | -0.3 (0.6) | -0.2 (0.7) | -1.1 (0.7)
  Erythema: Day 19 | -0.1 (0.7) | -0.3 (0.4) | -0.6 (0.8) | -0.5 (0.5) | -0.7 (0.6) | -1.4 (0.7)
  Scaling: Day 4 | 0.6 (0.7) | 0.6 (0.8) | -0.4 (0.6) | -0.3 (0.8) | -0.2 (0.5) | -1.3 (0.6)
  Scaling: Day 8 | 1.2 (0.8) | 1.1 (0.7) | -0.1 (0.5) | -0.2 (0.9) | -0.3 (1.0) | -1.3 (0.6)
  Scaling: Day 11 | 1.0 (1.0) | 1.0 (0.9) | -0.5 (0.8) | -0.3 (1.0) | -0.5 (1.0) | -1.7 (0.6)
  Scaling: Day 15 | 1.0 (1.0) | 0.9 (0.9) | -0.5 (0.8) | -0.3 (0.9) | -0.5 (0.7) | -1.5 (0.6)
  Scaling: Day 19 | 0.7 (1.0) | 0.4 (0.6) | -0.8 (0.8) | -0.8 (1.0) | -0.9 (0.6) | -1.8 (0.7)
  Induration: Day 4 | -0.0 (0.2) | -0.1 (0.3) | -0.0 (0.2) | -0.1 (0.3) | -0.0 (0.4) | -0.3 (0.5)
  Induration: Day 8 | 0.0 (0.3) | -0.1 (0.4) | 0.0 (0.3) | 0.0 (0.3) | -0.1 (0.4) | -0.4 (0.5)
  Induration: Day 11 | -0.2 (0.5) | -0.3 (0.6) | -0.4 (0.5) | -0.2 (0.4) | -0.3 (0.6) | -0.8 (0.4)
  Induration: Day 15 | -0.1 (0.6) | -0.2 (0.6) | -0.0 (0.6) | -0.0 (0.5) | -0.2 (0.5) | -0.8 (0.4)
  Induration: Day 19 | -0.4 (0.8) | -0.4 (0.6) | -0.3 (0.4) | -0.3 (0.5) | -0.3 (0.6) | -0.1 (0.5)

7. Secondary Outcome: Number of Participants With Success Rate at Each Visit
Description: Success rate was defined as a clearing score of 0 or 1, at each evaluation visit (Day 4, Day 8, Day 11, Day 15 and Day 19). The clearing score was ranged from 0 to 2, where scores were indicated as follows: 0=complete clearing (no scaling and no infiltration even on palpation. Post inflammatory hypo- or hyperpigmentation might be present, 1=almost clear (Residual erythema with some induration/infiltration [not clinically visible but palpable] without scaling, or residual erythema and residual scaling with no infiltration, 2=unchanged (unchanged or less than almost clear). Higher score indicated less success in clearing condition (worse outcome).
Time Frame: Day 4, Day 8, Day 11, Day 15 and Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Day 4: Yes | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: No | 24 | 24 | 24 | 24 | 24 | 24
  Day 8: Yes | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: No | 24 | 24 | 24 | 24 | 24 | 24
  Day 11: Yes | 0 | 0 | 0 | 0 | 0 | 5
  Day 11: No | 24 | 24 | 24 | 24 | 24 | 19
  Day 15: Yes | 1 | 0 | 0 | 0 | 0 | 2
  Day 15: No | 23 | 24 | 24 | 24 | 24 | 22
  Day 19: Yes | 1 | 1 | 0 | 1 | 1 | 7
  Day 19: No | 23 | 23 | 24 | 23 | 23 | 17

8. Secondary Outcome: Time to First Success
Description: The time to first success was defined as 0=no Success at any day, 1=success at Day 19 and not before, 2=success at Day 15 and not before, 3=success at Day 11 and not before, where lower score indicated less success in clearing condition (worse outcome).
Time Frame: Day 1 to Day 19
Population: Analysis was performed on ITT population, which comprised all participants who were randomized.
Measure: Count of Units; unit: mini-zones
Units Other Than Participants: mini-zones
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Number analyzed (mini-zones) | 24 | 24 | 24 | 24 | 24 | 24
mini-zones
  0-No success at any day | 23 | 23 | 24 | 23 | 23 | 15
  1-Success at Day 19 and not before | 0 | 1 | 0 | 1 | 1 | 4
  2-Success at Day 15 and not before | 1 | 0 | 0 | 0 | 0 | 0
  3-Success at Day 11 and not before | 0 | 0 | 0 | 0 | 0 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the informed consent form signature (up to 3 weeks before Day 1) until follow up (up to Day 26).
Description: Analysis was performed on safety population that included all participants who had received at least once the study treatment during the treatment period (from the day of first application of study treatment to the end of the study).
Groups:
- CD10367 Placebo Pretreated: Participants received 50 mcL matched placebo solution topically, on one or two desquamated psoriatic plaque (pre-treated), once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 3% Pretreated: Participants received 50 mcL 3% CD10367 solution topically, on one or two desquamated psoriatic plaque (pre-treated), once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 Placebo: Participants received matched placebo 50 mcL solution topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 1%: Participants received 50 mcL 1% CD10367 solution topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
- CD10367 3%: Participants received 50 mcL 3% CD10367 solution topically, on one or more psoriatic plaque, once daily, for 5 consecutive days a week for 2 weeks and 4 consecutive days in the third week.
Arm/Group | CD10367 Placebo Pretreated | CD10367 3% Pretreated | CD10367 Placebo | CD10367 1% | CD10367 3% | Betneval 0.1%
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 4/24 | 4/24 | 4/24 | 4/24 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD10367 Placebo Pretreated (N=24) | CD10367 3% Pretreated (N=24) | CD10367 Placebo (N=24) | CD10367 1% (N=24) | CD10367 3% (N=24) | Betneval 0.1% (N=24)
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 2 | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT03025282/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03025282/SAP_001.pdf